CLINICAL TRIAL: NCT05978193
Title: First-line Anti-PD-1 Therapy Plus Chemotherapy With or Without Radiotherapy in Metastatic Esophageal Squamous Cell Carcinoma: A Phase II Multi-center Trial (SCR-ESCC-01)
Brief Title: Radiotherapy Combined With Immunochemotherapy in Metastatic Esophageal Squamous Cell Carcinoma
Acronym: SCR-ESCC-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Wen Yu, Vice Director of Radiation Oncology Department, Shanghai Chest Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCR-ESCC-01
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Cancer; Metastatic Esophageal Squamous Cell Carcinoma
Keywords: Immunotherapy; low-dose radiotherapy; Esophageal squamous cell carcinoma; Immunoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Includes a single-arm safety run-in followed by randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): PD-1 inhibitor + Paclitaxel + Cisplatin/Carboplatin+ Low-dose radiotherapy (LDRT) + Conventionally fractionated radiotherapy (CFRT)
  Interventions: Radiation: LDRT+CFRT; Drug: Immunotherapy; Drug: Chemotherapy
- Arm B (Active Comparator): PD-1 inhibitor + Paclitaxel + Cisplatin/Carboplatin
  Interventions: Drug: Immunotherapy; Drug: Chemotherapy
- Safety Run-in Cohort (Experimental): Single Arm, LDRT + CFRT + Immunochemotherapy
  Interventions: Radiation: LDRT+CFRT; Drug: Immunotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: LDRT+CFRT — LDRT: Primary tumor and all visible metastatic lesions, DT: 2Gy/2fx, d1-2, Q3W × 4 cycles
  ; CFRT: Primary tumor, DT:40-50Gy/20-25fx, starting from the 5th immunotherapy cycle
  Arms: Arm A; Safety Run-in Cohort
Drug: Immunotherapy — PD-1 inhibitor 200mg, Q3W, until disease progression or unacceptable toxicity or treatment reaches 2 years
Drug: Chemotherapy — Paclitaxel+ Cisplatin, Q3W × 4cycles or Paclitaxel+ Carboplatin, Q3W × 4 cycles

SUMMARY:
SCR-ESCC-01 is a multicenter, randomized, phase II study aiming to investigate the benefit of early involvement of low-dose radiotherapy(LDRT) and conventionally fractionated radiotherapy(CFRT) in the first-line anti-PD-1 based treatment of metastatic ESCC. It begins with a safety run-in phase, followed by a randomized controlled comparison against standard immunochemotherapy.

DETAILED DESCRIPTION:
In metastatic esophageal squamous cell carcinoma (ESCC), radiotherapy is often administered for palliative purposes to alleviate dysphagia. Recent studies suggest that combining radiotherapy with immunotherapy may have a synergistic effect on treatment outcomes. This study aims to investigate the efficacy and safety of adding Low-Dose Radiotherapy (LDRT) combined with Conventionally Fractionated Radiotherapy (CFRT) to first-line immunochemotherapy.

Study Design:The protocol follows a sequential two-phase design:

1. Phase IIa (Safety Run-in / Pilot Phase):An initial cohort of approximately 20-25 patients will receive the experimental regimen (LDRT + CFRT + Immunochemotherapy) in a single-arm setting. The primary objective of this phase is to evaluate safety and feasibility.

   Safety Stopping Rule: A strict stopping rule is defined for the transition to the randomized phase. If 2 or more patients in the run-in cohort experience treatment-related death (Grade 5 Treatment-Related Adverse Events), the study will be terminated and will not proceed to Phase IIb.
2. Phase IIb (Randomized Controlled Phase):Upon confirmation that the safety criteria are met (i.e., < 2 treatment-related deaths and acceptable toxicity profile), subsequent patients will be randomly assigned (1:1) to:

Arm A (Experimental): PD-1 inhibitor plus chemotherapy (paclitaxel and platinum regimen) combined with LDRT and CFRT.

Arm B (Control): PD-1 inhibitor plus chemotherapy alone. Primary Endpoint:The primary endpoint for the randomized phase is median progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Metastatic esophageal squamous cell carcinoma (stage IVB, M1) confirmed by pathology;
3. ECOG performance status: 0-1 point;
4. No prior anti-tumor treatment;
5. Adequate hematologic, renal, hepatic, and cardiac functions that meet the requirements for chemotherapy and immunotherapy assessed by investigators.

Exclusion Criteria:

1. Non-squamous cell esophageal carcinoma or ESCC mixed with other pathological types of esophageal cancer;
2. Patients who are potentially curable with surgery as assessed by investigators;
3. Pleural metastasis or malignant pleural effusion, pericardial effusion;
4. Any prior anti-tumor therapy for esophageal cancer, i.e., surgery, radiotherapy, chemotherapy, or immunotherapy;
5. High risk of gastrointestinal bleeding, esophageal fistula, or perforation;
6. Patients with Patient-Generated Subjective Globe Assessment (PG-SGA) score≥9;
7. Unstable cardiac diseases or symptoms;
8. History of interstitial pulmonary disease, non-infectious pneumonitis; pulmonary fibrosis, or other uncontrolled acute pulmonary disease;
9. Active autoimmune disease or history of autoimmune disease;
10. Conditions of immunodeficiency or active infection requiring systemic therapy;
11. Pregnant or breastfeeding;
12. Patients with synchronous second primary cancer and a history of malignancy within the past 5 years (excluding completely cured cervical carcinoma in situ or basal cell or squamous cell skin carcinoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival
Safety and Feasibility of the Combined Regimen (Safety Run-in Phase) | From start of treatment up to 30 days after the last dose.
  Incidence of Treatment-Related Adverse Events (TRAEs) in the initial cohort.

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 36 months
  Median overall survival
Incidence of Grade III and higher treatment-related adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wen Yu, M.D, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Shanghai Ruijin Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] Lu Z, Wang J, Shu Y, Liu L, Kong L, Yang L, Wang B, Sun G, Ji Y, Cao G, Liu H, Cui T, Li N, Qiu W, Li G, Hou X, Luo H, Xue L, Zhang Y, Yue W, Liu Z, Wang X, Gao S, Pan Y, Galais MP, Zaanan A, Ma Z, Li H, Wang Y, Shen L; ORIENT-15 study group. Sintilimab versus placebo in combination with chemotherapy as first line treatment for locally advanced or metastatic oesophageal squamous cell carcinoma (ORIENT-15): multicentre, randomised, double blind, phase 3 trial. BMJ. 2022 Apr 19;377:e068714. doi: 10.1136/bmj-2021-068714. PMID 35440464
- [Background] Wang ZX, Cui C, Yao J, Zhang Y, Li M, Feng J, Yang S, Fan Y, Shi J, Zhang X, Shen L, Shu Y, Wang C, Dai T, Mao T, Chen L, Guo Z, Liu B, Pan H, Cang S, Jiang Y, Wang J, Ye M, Chen Z, Jiang D, Lin Q, Ren W, Wang J, Wu L, Xu Y, Miao Z, Sun M, Xie C, Liu Y, Wang Q, Zhao L, Li Q, Huang C, Jiang K, Yang K, Li D, Liu Y, Zhu Z, Chen R, Jia L, Li W, Liao W, Liu HX, Ma D, Ma J, Qin Y, Shi Z, Wei Q, Xiao K, Zhang Y, Zhang Y, Chen X, Dai G, He J, Li J, Li G, Liu Y, Liu Z, Yuan X, Zhang J, Fu Z, He Y, Ju F, Liu Z, Tang P, Wang T, Wang W, Zhang J, Luo X, Tang X, May R, Feng H, Yao S, Keegan P, Xu RH, Wang F. Toripalimab plus chemotherapy in treatment-naive, advanced esophageal squamous cell carcinoma (JUPITER-06): A multi-center phase 3 trial. Cancer Cell. 2022 Mar 14;40(3):277-288.e3. doi: 10.1016/j.ccell.2022.02.007. Epub 2022 Mar 3. PMID 35245446
- [Background] Herrera FG, Bourhis J, Coukos G. Radiotherapy combination opportunities leveraging immunity for the next oncology practice. CA Cancer J Clin. 2017 Jan;67(1):65-85. doi: 10.3322/caac.21358. Epub 2016 Aug 29. PMID 27570942
- [Background] Shaverdian N, Lisberg AE, Bornazyan K, Veruttipong D, Goldman JW, Formenti SC, Garon EB, Lee P. Previous radiotherapy and the clinical activity and toxicity of pembrolizumab in the treatment of non-small-cell lung cancer: a secondary analysis of the KEYNOTE-001 phase 1 trial. Lancet Oncol. 2017 Jul;18(7):895-903. doi: 10.1016/S1470-2045(17)30380-7. Epub 2017 May 24. PMID 28551359
- [Background] Theelen WSME, Peulen HMU, Lalezari F, van der Noort V, de Vries JF, Aerts JGJV, Dumoulin DW, Bahce I, Niemeijer AN, de Langen AJ, Monkhorst K, Baas P. Effect of Pembrolizumab After Stereotactic Body Radiotherapy vs Pembrolizumab Alone on Tumor Response in Patients With Advanced Non-Small Cell Lung Cancer: Results of the PEMBRO-RT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1276-1282. doi: 10.1001/jamaoncol.2019.1478. PMID 31294749
- [Background] Herrera FG, Ronet C, Ochoa de Olza M, Barras D, Crespo I, Andreatta M, Corria-Osorio J, Spill A, Benedetti F, Genolet R, Orcurto A, Imbimbo M, Ghisoni E, Navarro Rodrigo B, Berthold DR, Sarivalasis A, Zaman K, Duran R, Dromain C, Prior J, Schaefer N, Bourhis J, Dimopoulou G, Tsourti Z, Messemaker M, Smith T, Warren SE, Foukas P, Rusakiewicz S, Pittet MJ, Zimmermann S, Sempoux C, Dafni U, Harari A, Kandalaft LE, Carmona SJ, Dangaj Laniti D, Irving M, Coukos G. Low-Dose Radiotherapy Reverses Tumor Immune Desertification and Resistance to Immunotherapy. Cancer Discov. 2022 Jan;12(1):108-133. doi: 10.1158/2159-8290.CD-21-0003. Epub 2021 Sep 3. PMID 34479871
- [Background] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411
- [Derived] Li Y, Lin L, Liu J, Cai XW, Zhang Q, Song XY, Zhao SG, Ma XM, Fu XL, Yu W. Phase II multicenter trial: first-line immunochemotherapy with or without radiotherapy in metastatic esophageal squamous cell cancer (SCR-ESCC-01). Future Oncol. 2023 Nov;19(34):2291-2296. doi: 10.2217/fon-2023-0674. Epub 2023 Nov 8. PMID 37937444